CLINICAL TRIAL: NCT03606733
Title: Suprachoroidal Injection of Triamcinolone Acetonide Using Custom Made Needle to Treat Macular Diseases and Non Infectious Posterior Uveitis
Brief Title: Suprachoroidal Injection of Triamcinolone Acetonide Using Custom Made Needle to Treat Retinal Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Marashi Eye Clinic (Other)
Responsible Party: Principal Investigator, Ameen Marashi, Principle investigator, Marashi Eye Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCS
Record Dates: First submitted 2018-07-22; First posted 2018-07-31 (Actual); Last update posted 2018-10-29 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Macular Edema, Cystoid Macular Edema, Chorodial Neovascularzation, Posterior Uveitis
MeSH Terms: conditions — Macular Edema; Uveitis, Posterior

STUDY DESIGN:
Intervention Model Description: Injection of triamcinilone or/ and VEGF blockade agents in the Supra Choroidal Space
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- A custom made Suprachoroidal needle for macular diseases (Experimental): A custom made 30 gauge needle offering 1000 micron penetration of the sclera at the parsplana
  Interventions: Procedure: Custom suorachoroidal needle

INTERVENTIONS:
Procedure: Custom suorachoroidal needle — Custom made Supra Choroidal Space needle

SUMMARY:
Injection in the Suprachoroidal space has potential of increasing the efficacy of the drug upto six times with direct effect on retinal tissues sparing the crystalline lens and trabecular meshwork.

DETAILED DESCRIPTION:
A custom made 30 gauge needle offering 1000 micron penetration of the sclera at the parsplana with the help of gentle pressure on the sclera will help to inject medication such as triamcinilone or VEGF blockade agents (Ziv aflibercept or Bevacizumab) in the potential Suprachoroidal space which offers direct effect of injected drug on the retina and choroid sparing both crystalline lens, trabecular meshwork and other ocular tissues, hence improving efficacy of the drug upto six times and reduce potential complications such as cataract and glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* 20 years and older
* Patients with macular edema or degeneration from various pathologies
* Central macular thickness more than 250 microns
* Patients who are able to come for all follow-up

Exclusion Criteria:

* Significant renal disease, defined as a history of chronic renal failure requiring dialysis or kidney transplant.
* Myocardial infarction, other acute cardiac event requiring hospitalization, stroke, transient ischemic attack, or treatment for acute congestive heart failure within 4 months prior to randomization
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 3 years.
* Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-08-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients achieved visual acuity improvement | 12 weeks
  To measure best corrected visual acuity using using Snellen chart or equivalent

SECONDARY OUTCOMES:
Amount of Central macular thickness reduction in microns | 12 weeks
  Using optical coherence tomography in monthly bases to measure central retinal thickness
Proportion of eyes with Increased intraocular pressure | 12 weeks
  To measure intraocular pressure using Goldmann applanation tonometer

CONTACTS AND LOCATIONS:
Locations (1):
- Marashi Eye Clinic, Aleppo, Syria

REFERENCES:
- [Background] Marashi A. Treating macular edema secondary to retinal vein occlusion with suprachoroidal injection of triamcinolone acetonide using custom made needle. Adv Ophthalmol Vis Syst. 2018;8(5):277-281. DOI: 10.15406/aovs.2018.08.00321
- See also: Treating macular edema secondary to retinal vein occlusion with suprachoroidal injection of triamcinolone acetonide using custom made needle — http://medcraveonline.com/AOVS/AOVS-08-00321.pdf